CLINICAL TRIAL: NCT00006483
Title: A Phase II Study Of Aerosolized GM-CSF In The Treatment Of Metastatic Renal Cell Carcinoma To The Lung
Brief Title: Sargramostim in Treating Patients With Kidney Cancer That Has Spread to the Lung
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N9953; CDR0000068314 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2000-11-06; First posted 2004-04-29 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Kidney Cancer; Metastatic Cancer
Keywords: stage IV renal cell cancer; recurrent renal cell cancer; lung metastases
MeSH Terms: conditions — Kidney Neoplasms; Neoplasm Metastasis; Carcinoma, Renal Cell | interventions — sargramostim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- aerosolized sargramostim (Experimental): Patients receive aerosolized sargramostim (GM-CSF) by nebulizer over 10-15 minutes twice daily on days 1-7 and 14-21. Treatment repeats every 28 days in the absence of disease progression or unaceptable toxicity.
  Patients are followed for disease progression and then every 3 months thereafter.
  Interventions: Biological: sargramostim

INTERVENTIONS:
Biological: sargramostim

SUMMARY:
RATIONALE: Colony-stimulating factors such as sargramostim may increase the number of immune cells found in bone marrow or peripheral blood and may be an effective treatment for patients with kidney cancer that has spread to the lung.

PURPOSE: Phase II trial to study the effectiveness of sargramostim in treating patients who have kidney cancer that has spread to the lung.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the 4-month progression-free survival rate and overall survival rate in patients with metastatic renal cell carcinoma to the lung treated with aerosolized sargramostim (GM-CSF).
* Determine the toxicity of this regimen in these patients.
* Determine the immunomodulatory effects of this regimen in terms of natural killer cells cytotoxicity, and T-cell, B-cell, and dendritic cell activation markers.

OUTLINE: This is a multicenter study.

Patients receive aerosolized sargramostim (GM-CSF) by nebulizer over 10-15 minutes twice daily on days 1-7 and 14-21. Treatment repeats every 28 days in the absence of disease progression or unaceptable toxicity.

Patients are followed for disease progression and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 21-48 patients will be accrued for this study within 7-20 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic renal cell carcinoma for which no known standard therapy that is potentially curative or capable of extending life expectancy exists (e.g., surgery)
* Measurable metastatic disease in the lung

  * At least one unidimensionally measurable lesion at least 20 mm by conventional techniques
* No CNS metastases that require treatment

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 12 weeks

Hematopoietic

* Absolute neutrophil count at least 1,000/mm^3
* Platelet count at least 75,000/mm^3
* Hemoglobin greater than 8.0 g/dL

Hepatic

* Bilirubin no greater than 2 times upper limit of normal (ULN)
* AST no greater than 3 times ULN

Renal

* Creatinine no greater than 2.5 times ULN

Pulmonary

* No hemoptysis of grade 3 or greater
* No reactive airway disease on active therapy

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No uncontrolled infection
* No other metastatic malignancy within the past 3 years except basal cell skin cancer

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 2 weeks since prior immunotherapy
* More than 2 weeks since other prior biologic therapy

Chemotherapy

* More than 3 weeks since prior chemotherapy (6 weeks for mitomycin or nitrosoureas)

Endocrine therapy

* More than 2 weeks since prior corticosteroids
* No concurrent systemic glucocorticoids

Radiotherapy

* More than 2 weeks since prior radiotherapy
* No prior radiotherapy to more than 10% of total lung volume in the radiation field

Other

* At least 4 weeks since prior bronchodialators
* No concurrent immunosuppressive agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2000-10; Primary Completion 2003-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Determine the 4-month progression-free survival rate | 4 months

SECONDARY OUTCOMES:
Determine the 4-month overall survival rate | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Svetomir Markovic, MD, PhD, Study Chair — Mayo Clinic
Locations (24):
- United States (22):
  - CCOP - Scottsdale Oncology Program, Scottsdale, Arizona
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Ochsner, New Orleans, Louisiana
  - CCOP - Ann Arbor Regional, Ann Arbor, Michigan
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CentraCare Clinic, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - CCOP - Missouri Valley Cancer Consortium, Omaha, Nebraska
  - Quain & Ramstad Clinic, P.C., Bismarck, North Dakota
  - CCOP - Merit Care Hospital, Fargo, North Dakota
  - Altru Health Systems, Grand Forks, North Dakota
  - CCOP - Toledo Community Hospital Oncology Program, Toledo, Ohio
  - CCOP - Geisinger Clinic and Medical Center, Danville, Pennsylvania
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota
  - Central Plains Clinic, Ltd., Sioux Falls, South Dakota
- Canada (2):
  - Saskatchewan Cancer Agency, Regina, Saskatchewan
  - Allan Blair Cancer Centre, Regina, Saskatchewan